CLINICAL TRIAL: NCT00003146
Title: A Phase II Trial of Thiotepa, Busulfan, and Melphalan Followed by Autologous or Syngeneic Marrow or Peripheral Blood Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Combination Chemotherapy Followed by Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1204.00; FHCRC-1204.00; NCI-H97-0007; CDR0000065929 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Busulfan; Melphalan; Thiotepa; Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: busulfan
Drug: melphalan
Drug: thiotepa
Procedure: bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by bone marrow or peripheral stem cell transplantation in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity and efficacy at the maximum tolerated dose of busulfan, melphalan, and thiotepa in patients with multiple myeloma.

OUTLINE: This is a single arm, open label study. Peripheral blood stem cells (PBSC) are collected and cryopreserved, or bone marrow is harvested and stored, until infusion on day 0. Patients receive oral busulfan every 6 hours on days -8, -7, and -6. Melphalan is administered by continuous IV infusion over 30 minutes on days -5 and -4. Thiotepa is administered by continuous IV infusion over 2 hours on days -3 and -2. Patients undergo PBSC or bone marrow infusion 36-48 hours following the completion of chemotherapy (day 0). Patients are followed for 100 days posttransplant and every 3 months thereafter.

PROJECTED ACCRUAL: 30 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed stage II/III multiple myeloma (or have greater than normal beta-2-microglobulin) meeting the Salmon and Durie criteria Stage I multiple myeloma must have had prior chemotherapy before undergoing transplantation

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine clearance at least 50 mg/min Cardiovascular: Left ventricular ejection fraction at least 41% Other: Not pregnant HIV negative

PRIOR CONCURRENT THERAPY: Not specified

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-11; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States